CLINICAL TRIAL: NCT04587271
Title: Investigating the Impact of Moringa Oleifera Leaf Supplementation on Growth, Nutrition, Lactation, and Inflammation in Kenyan Breastfeeding Mothers and Children
Brief Title: Nutritional Impact of Moringa Oleifera Leaf Supplementation in Mothers and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzanna L Attia (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor-Investigator, Suzanna L Attia, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 58219; K01TW009987-06 (NIH)
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-10

CONDITIONS: Malnutrition; Wasting; Growth Failure
Keywords: Moringa oleifera; supplementation
MeSH Terms: conditions — Malnutrition; Cachexia; Failure to Thrive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Lactating Mothers (Moringa) (Experimental): Lactating mothers.
  Interventions: Dietary Supplement: Moringa oleifera (high dose)
- Breastfeeding Infants (Moringa) (Experimental): Breastfeeding infants from lactating mothers
  Interventions: Dietary Supplement: Moringa oleifera (high dose)
- Children (Moringa) (Experimental): Children from 6-59 months of age.
  Interventions: Dietary Supplement: Moringa oleifera (low dose)
- Lactating Mothers (placebo) (Placebo Comparator): Lactating mothers.
  Interventions: Dietary Supplement: Placebo
- Breastfeeding Infants (placebo) (Placebo Comparator): Breastfeeding infants from lactating mothers
  Interventions: Dietary Supplement: Placebo
- Children (placebo) (Placebo Comparator): Children from 6-59 months of age.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Moringa oleifera (high dose) — Mothers will receive 20 grams of moringa leaf powder in porridge consumed daily for three months.
  Arms: Breastfeeding Infants (Moringa); Lactating Mothers (Moringa)
Dietary Supplement: Moringa oleifera (low dose) — Children will receive 5-10 grams of moringa leaf powder in porridge consumed daily for three months.
  Arms: Children (Moringa)
Dietary Supplement: Placebo — Mothers and children will receive porridge with placebo.
  Arms: Breastfeeding Infants (placebo); Children (placebo); Lactating Mothers (placebo)

SUMMARY:
Studies to date on the effects of Moringa oleifera in diabetes and anemia and animal studies that examine the utility of moringa for increased milk and litter yield are of small scale, however high-quality large-scale placebo or case-controlled clinical trials to define the impact on infants of moringa leaf powder consumption by breastfeeding mothers are lacking. Moringa has a traditional and agricultural history of use as a galactagogue; despite this and its incorporation into products such as Mother's Milk Tea© and placement on NIH LactMed Lactation Database, this property has not been studied in large clinical trials nor in populations dependent on breastmilk such as in Kisumu, Kenya. This study will improve and add to existing knowledge of moringa's effect on human breastmilk and will provide novel information on the effect of moringa supplementation to lactating mothers on their infant's intestinal inflammation and health. After trial registration, the study was modified to include infant follow up to 18 months for some measures and the children's groups were removed. Although the study was modified to an 18 month follow up, the data were not able to be collected.

Further understanding of the acceptability of moringa leaf in a staple food of porridge and more the effect of moringa supplementation on infant and childhood growth, nutrition, and intestinal and systemic inflammation may translate in the future to the cultivation of moringa at the community or household level as an effective resource for the improvement of childhood undernutrition.

ELIGIBILITY:
Inclusion Criteria:

* lactating women at least 18 years of age and their exclusively breastfed infants within 14 days of delivery.
* children 6-59 months of age who eat food

Exclusion Criteria:

* regular maternal consumption of moringa
* receipt and consumption of food supplementation program
* inability to feed orally or refusal to eat moringa or placebo porridge
* for infants, prematurity (<36 weeks gestational age)
* for infants, significant congenital disease
* for infants, inability to feed orally

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2022-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna L Attia, Principal Investigator — University of Kentucky
Locations (2):
- Kenya (2):
  - Kombewa County Hospital, Kisumu
  - Chulaimbo Sub- County Hospital, Kisumu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Attia SL, Owuor PM, Odhiambo SA, Mogaka JN, Ondondo R, Navarro IC, Schadler A, McQuerry K, Fuchs GJ 3rd, Williams JE, Scarrow KN, McGuire MA, McGuire MK, Waterman C. Effect of Maternal Moringa oleifera Leaf Supplementation on Maternal and Infant Nutritional Status and Human Milk Output: A Pilot Single-Blinded Cluster-Randomized Trial. Curr Dev Nutr. 2025 Oct 3;9(11):107568. doi: 10.1016/j.cdnut.2025.107568. eCollection 2025 Nov. PMID 41282517

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After trial registration, the children's groups were removed so no children were enrolled in the study
Period: Overall Study
Arm/Group | Lactating Mothers (Moringa) | Breastfeeding Infants (Moringa) | Children (Moringa) | Lactating Mothers (Placebo) | Breastfeeding Infants (Placebo) | Children (Placebo)
Started | 25 | 25 | 0 | 25 | 25 | 0
Completed | 23 | 23 | 0 | 22 | 23 | 0
Not Completed | 2 | 2 | 0 | 3 | 2 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0 | 2 | 2 | 0
Not completed — Caregiver brought child to visits | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactating Mothers (Moringa) | Breastfeeding Infants (Moringa) | Lactating Mothers (Placebo) | Breastfeeding Infants (Placebo) | Total
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] — Totals include combined data from mothers and infants
  years | 27.2 (6) | 0.04 (0.02) | 27.8 (6.2) | .05 (.02) | 13.8 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 9 | 25 | 13 | 72
  Male | 0 | 16 | 0 | 12 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 25 | 25 | 25 | 25 | 100
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 25 | 25 | 25 | 25 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Body weight
Time Frame: at baseline and 3 months
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Lactating Mothers (Moringa) | Breastfeeding Infants (Moringa) | Lactating Mothers (Placebo) | Breastfeeding Infants (Placebo)
Number analyzed (Participants) | 23 | 23 | 22 | 23
g | 365 (3102) | 2.5 (0.9) | -470 (2988) | 2.5 (0.8)

2. Secondary Outcome: Change in Infant Height
Description: Height (body length)
Time Frame: at baseline and 3 months
Population: Height was not measured in the mothers
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Breastfeeding Infants (Moringa) | Breastfeeding Infants (Placebo)
Number analyzed (Participants) | 23 | 23
cm | 9.1 (2.1) | 9.3 (1.7)

3. Secondary Outcome: Change in Mid-Upper Arm Circumference
Description: Mid-upper arm circumference (MUAC) will be measured at baseline and monthly to 3 months. Change from baseline to 3 months reported
Time Frame: baseline and 3 months
Population: change in MUAC was not measured in the infants
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Lactating Mothers (Moringa) | Lactating Mothers (Placebo)
Number analyzed (Participants) | 23 | 22
cm | -1.7 (1.5) | -1.6 (1.5)

4. Secondary Outcome: Change in Vitamin A
Description: Serum retinol binding protein will be used to survey vitamin A levels in infants at baseline and monthly to 3 months..
Time Frame: 3 months
Population: 1 additional participant in the placebo group of mothers provided blood work (23 total as opposed to 22 from the participant flow section); Unable to get blood samples from 1 pair in the Moringa group (22 total as opposed to 23 from the participant flow section)
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Lactating Mothers (Moringa) | Breastfeeding Infants (Moringa) | Lactating Mothers (Placebo) | Breastfeeding Infants (Placebo)
Number analyzed (Participants) | 22 | 22 | 23 | 23
mcmol/L | -0.29 (0.50) | 0.08 (0.48) | -0.23 (0.69) | 0.09 (0.50)

5. Secondary Outcome: Change in CRP Levels
Description: C-reactive protein (CRP) will be used to measure inflammation at baseline and monthly to 3 months. Change from baseline to 3 months reported. Negative values are considered a better outcome.
Time Frame: baseline and 3 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Lactating Mothers (Moringa) | Breastfeeding Infants (Moringa) | Lactating Mothers (Placebo) | Breastfeeding Infants (Placebo)
Number analyzed (Participants) | 22 | 22 | 23 | 23
mg/L | -3.5 (11.6) | 2.3 (6.3) | -5.3 (8.1) | 8.8 (18.7)

6. Secondary Outcome: Change in the Soluble Transferrin Receptor
Description: The soluble transferrin receptor (sTFR) will be used to evaluate anemia at baseline and monthly to 3 months. Change from baseline to 3 months reported.
Time Frame: baseline and 3 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Lactating Mothers (Moringa) | Breastfeeding Infants (Moringa) | Lactating Mothers (Placebo) | Breastfeeding Infants (Placebo)
Number analyzed (Participants) | 22 | 22 | 23 | 23
mg/L | -0.1 (2.8) | 2.5 (2.1) | -1.3 (2.6) | 1.8 (2.7)

7. Secondary Outcome: Change in Fecal Neopterin
Description: Fecal neopterin will be measured at baseline and at 3 months.
Time Frame: baseline and 3 months
Population: 21 stool samples for the moringa group and 22 for the placebo group were successfully analyzed for mothers and infants.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Lactating Mothers (Moringa) | Breastfeeding Infants (Moringa) | Lactating Mothers (Placebo) | Breastfeeding Infants (Placebo)
Number analyzed (Participants) | 21 | 21 | 22 | 22
nmol/L | 21.56 (39.05) | 1076.44 (1387.85) | 26.09 (49.42) | 791.08 (868.18)

8. Secondary Outcome: Change in Fecal Myeloperoxidase
Description: Fecal myeloperoxidase will be measured at baseline and at 3 months.
Time Frame: baseline and 3 months
Population: 21 stool samples for the moringa group and 22 for the placebo group were successfully analyzed for mothers and infants.
Measure: Mean (Standard Deviation); unit: ng/ML
Arm/Group | Lactating Mothers (Moringa) | Breastfeeding Infants (Moringa) | Lactating Mothers (Placebo) | Breastfeeding Infants (Placebo)
Number analyzed (Participants) | 21 | 21 | 22 | 22
ng/ML | 35.93 (682.23) | 1071.01 (2687.39) | 105.02 (348.27) | 1225.78 (1276.9)

9. Secondary Outcome: Change in Alpha-1-Antitrypsin
Description: Fecal alpha-1-antitrypsin will be measured at baseline and at 3 months.
Time Frame: baseline and 3 months
Population: 21 stool samples for the moringa group and 22 for the placebo group were successfully analyzed for mothers and infants.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Lactating Mothers (Moringa) | Breastfeeding Infants (Moringa) | Lactating Mothers (Placebo) | Breastfeeding Infants (Placebo)
Number analyzed (Participants) | 21 | 21 | 22 | 22
mcg/L | 3.28 (25.57) | -29.12 (195.56) | 0.61 (6.49) | 66.04 (125.94)

10. Secondary Outcome: Change in the Prevalence of Diarrhea
Description: Proportion of participants experiencing diarrhea (> 3 watery stools in 24 hours).
Time Frame: 1 and 3 months
Measure: Number; unit: participants
Arm/Group | Lactating Mothers (Moringa) | Breastfeeding Infants (Moringa) | Lactating Mothers (Placebo) | Breastfeeding Infants (Placebo)
Number analyzed (Participants) | 23 | 23 | 22 | 23
participants | -2 | 1 | -1 | 3

11. Secondary Outcome: Change in Breastmilk Volume
Description: Breastmilk volume will be assessed from 24 hour breast pumping or hand expression or weighing the infant before and after feeding for 24 hours.
Time Frame: at enrollment and at 3 months
Population: unable to review 24-hour pumped information from 1 mother in the placebo group
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Lactating Mothers (Moringa) | Lactating Mothers (Placebo)
Number analyzed (Participants) | 23 | 21
mL | 435.9 (381.5) | 12.4 (465.7)

12. Secondary Outcome: Change in Breastmilk Vitamin A
Description: Levels of vitamin A in breastmilk will be measured at the end of the study.
Time Frame: baseline and 3 months
Population: outcome measure data not reported because unable to perform vitamin A analysis due to funding limitations
Arm/Group | Lactating Mothers (Moringa) | Lactating Mothers (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Diarrhea is a common occurrence in this region (Western Kenya) due to a high prevalence of parasitic, viral, and bacterial infections. Therefore diarrhea is not considered an adverse event in this study.
Arm/Group | Lactating Mothers (Moringa) | Breastfeeding Infants (Moringa) | Lactating Mothers (Placebo) | Breastfeeding Infants (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT04587271/Prot_SAP_ICF_001.pdf